CLINICAL TRIAL: NCT04376528
Title: Mycophenolate Mofetil Versus Cyclosporin A in the Treatment of Primary Biliary Cholangitis-autoimmune Hepatitis Overlap Syndrome Duo to Nonresponse to Standard Therapy
Brief Title: Mycophenolate Mofetil Versus Cyclosporin A in the Treatment of Primary Biliary Cholangitis-autoimmune Hepatitis Overlap Syndrome Due to Nonresponse to Standard Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Li Yang, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OS-3
Record Dates: First submitted 2020-05-03; First posted 2020-05-06 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-05

CONDITIONS: Hepatitis, Autoimmune; Primary Biliary Cholangitis; Immunosuppression
MeSH Terms: conditions — Hepatitis, Autoimmune; Liver Cirrhosis, Biliary | interventions — Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclosporin A (Experimental)
  Interventions: Drug: Cyclosporin A
- Mycophenolate Mofetil (Active Comparator)
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Cyclosporin A — Ursodeoxycholic acid combination of immunosuppressive agents(methylprednisolone with cyclosporin A)
  Arms: Cyclosporin A
Drug: Mycophenolate Mofetil — Ursodeoxycholic acid combination of immunosuppressive agents(methylprednisolone with mycophenolate mofetil )
  Arms: Mycophenolate Mofetil

SUMMARY:
Biochemical response of primary biliary cholangitis-autoimmune hepatitis overlap syndrome induced by mycophenolate mofetil versus cyclosporin A

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-70 years;
2. Diagnosed with PBC-AIH overlap syndrome according to Paris criteria;
3. Patients have a nonresponse to azathioprine;
4. The WBC count ≥2.5x10^9/L and platelet count ≥50x10^9/L.
5. Agreed to participate in the trial, and assigned informed consent;

Exclusion Criteria:

1. The presence of hepatitis A, B, C, D, or E virus infection;
2. Patients with presence of serious decompensated cirrhosis;
3. Patients have a history of glucocorticoid or immunosuppressant medication before enrollment;
4. Liver damage caused by other reasons: such as primary sclerosing cholangitis, non-alcoholic steatohepatitis, drug induced liver disease or Wilson's disease.
5. Pregnant and breeding women and women of childbearing age in need of reproduction
6. Severe disorders of other vital organs, such as severe heart failure, cancer;
7. Patients with presence of renal insufficiency;
8. Parenteral administration of blood or blood products within 6 months before screening;
9. Recent treatment with drugs having known liver toxicity;
10. Taken part in other clinic trials within 6 months before enrollment.
11. Patients who are allergic to these drugs;
12. Uncontrolled infection and hypertension ;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Biochemical remission | up to 6 months
  The percentage of patients in biochemical remission, defined as normalization of serum ALT and IgG levels after 24 weeks of treatment, per treatment group.

SECONDARY OUTCOMES:
Partial remission | up to 6 months
  Partial remission, defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) serum levels >1x Upper Limit of Normal (ULN) and <2x ULN
Minimal response | up to 6 months
  Minimal response, defined as decrease of ALT or AST serum levels but still >2x ULN
Treatment failure | up to 6 months
  defined as no improvement or increase of ALT or AST serum levels
Changes in liver stiffness | up to 6 months
  liver stiffness will be measured by shear-wave elastography
Side-effects | up to 6 months
  Drug related side-effects

CONTACTS AND LOCATIONS:
Locations (1):
- WestChina Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No